CLINICAL TRIAL: NCT02341066
Title: Evaluation of a New Score Incorporating Endothelial Dysfunction for the Assessment of Coronary Heart Disease Risk in Patients With Rheumatoid Arthritis: a 3-year Prospective Study.
Brief Title: Endothelial Dysfunction Evaluation for Coronary Heart Disease Risk Estimation in Rheumatoid Arthritis (EDRA Study)
Acronym: EDRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria di Sassari (Other)
Collaborators: Azienda Ospedaliero Universitaria di Cagliari (Other); Complesso Integrato Columbus, Roma (Unknown)
Responsible Party: Principal Investigator, Gian Luca Erre, MD PhD, MD, PhD, Azienda Ospedaliero Universitaria di Sassari
Other Study IDs: H89D14000850003; GR-2011-02352816 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis; Coronary Heart Disease
Keywords: Cardiovascular risk score; Framingham risk score 2-year; Endothelial dysfunction; EndoPAT; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis: Rheumatoid arthritis patients free of overt cardiovascular disease. Endothelial Dysfunction evaluation by EndoPAT
  Interventions: Device: Endothelial Dysfunction evaluation by EndoPAT

INTERVENTIONS:
Device: Endothelial Dysfunction evaluation by EndoPAT — Endothelial dysfunction will be measured assessing reactive hyperemia of digital arteries by using Endo-PAT2000 (Itamar, Israel).

SUMMARY:
To evaluate the contribution of the assessment of endothelial dysfunction (ED) in improving coronary hearth disease (CHD) risk stratification obtained by the Framingham risk score (FRS) in rheumatoid arthritis population (RA).

DETAILED DESCRIPTION:
ED, determined by peripheral arterial tonometry (PAT), will be evaluated at baseline in 3000 RA patients free of previous cardiovascular events. Incident CHD events during the 3-year planned follow-up will be registered. A measure of the incremental yield of ED will be obtained comparing 2-year Framingham risk score for CHD (FRS) and FRS plus ED differential prognostic performances by C-statics and risk reclassification analysis.

ELIGIBILITY:
Inclusion Criteria:

* RA as defined by American College of Rheumatology/European League Against Rheumatisms 2010 RA classification criteria
* In the opinion of investigators, patients must be able to adhere to the study visit schedule and must be capable of giving informed consent

Exclusion Criteria:

* Previous cardiovascular or cerebrovascular events (acute coronary syndrome, stable angina, stroke, interventional procedures, carotid endarterectomy, symptomatic peripheral artery ischemia)
* Pathological ECG at rest
* Sign or symptoms of autonomous nervous system dysfunction
* Serious infections in the previous 6 months
* Concomitant severe illness: overt hepatic insufficiency; End stage renal disease (Glomerular Filtration Rate <30 ml/h at Cockrofts-Gault formula); recent diagnosis of cancer
* Pregnancy
* Plans to leave target areas of each study site within three years

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three thousand consecutive RA patients free of overt cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
CHD events | 3 year
  The following events will be considered as incident CHD events: myocardial infarction, CHD death, resuscitated cardiac arrest, or definite or probable angina if followed by coronary revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Erre, MD, PhD, Principal Investigator — Azienda Ospedaliero Universitaria di Sassari
Locations (3):
- Italy (3):
  - Policlinico Universitario di Monserrato Azienda Ospedaliera Universitaria di Cagliari, Monserrato, Cagliari
  - Complesso Integrato Columbus, UO di Reumatologia, Roma, Roma
  - Azienda Ospedaliero Universitaria di Sassari, UOC di Reumatologia, Sassari, Sassari

REFERENCES:
- [Background] D'Agostino RB, Russell MW, Huse DM, Ellison RC, Silbershatz H, Wilson PW, Hartz SC. Primary and subsequent coronary risk appraisal: new results from the Framingham study. Am Heart J. 2000 Feb;139(2 Pt 1):272-81. doi: 10.1067/mhj.2000.96469. PMID 10650300
- [Background] Crowson CS, Matteson EL, Roger VL, Therneau TM, Gabriel SE. Usefulness of risk scores to estimate the risk of cardiovascular disease in patients with rheumatoid arthritis. Am J Cardiol. 2012 Aug 1;110(3):420-4. doi: 10.1016/j.amjcard.2012.03.044. Epub 2012 Apr 20. PMID 22521305
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Matsuzawa Y, Sugiyama S, Sugamura K, Nozaki T, Ohba K, Konishi M, Matsubara J, Sumida H, Kaikita K, Kojima S, Nagayoshi Y, Yamamuro M, Izumiya Y, Iwashita S, Matsui K, Jinnouchi H, Kimura K, Umemura S, Ogawa H. Digital assessment of endothelial function and ischemic heart disease in women. J Am Coll Cardiol. 2010 Apr 20;55(16):1688-96. doi: 10.1016/j.jacc.2009.10.073. PMID 20394872
- [Background] Rubinshtein R, Kuvin JT, Soffler M, Lennon RJ, Lavi S, Nelson RE, Pumper GM, Lerman LO, Lerman A. Assessment of endothelial function by non-invasive peripheral arterial tonometry predicts late cardiovascular adverse events. Eur Heart J. 2010 May;31(9):1142-8. doi: 10.1093/eurheartj/ehq010. Epub 2010 Feb 24. PMID 20181680
- [Derived] Erre GL, Chessa I, Bassu S, Cavagna L, Carru C, Pintus G, Giordo R, Mangoni AA, Damiano Sanna G, Zinellu A. Association between ischemia-modified albumin (IMA) and peripheral endothelial dysfunction in rheumatoid arthritis patients. Sci Rep. 2024 Feb 17;14(1):3964. doi: 10.1038/s41598-024-54641-5. PMID 38368495
- [Derived] Sanna GD, Piga M, Piga A, Falco O, Ponti E, Cauli A, Floris A, Mangoni AA, Casu G, De Luca G, Erre GL; EDRA Study Group. Prevalence and clinical significance of electrocardiographic signs of atrial myopathy in rheumatoid arthritis: results from the EDRA study. Clin Exp Rheumatol. 2023 Jul;41(7):1427-1433. doi: 10.55563/clinexprheumatol/d9l4lt. Epub 2023 Jan 2. PMID 36622121
- [Derived] Erre GL, Mangoni AA, Passiu G, Bassu S, Castagna F, Carru C, Piga M, Zinellu A, Sotgia S. Comprehensive arginine metabolomics and peripheral vasodilatory capacity in rheumatoid arthritis: A monocentric cross-sectional study. Microvasc Res. 2020 Sep;131:104038. doi: 10.1016/j.mvr.2020.104038. Epub 2020 Jul 2. PMID 32622695
- [Derived] Erre GL, Ferraccioli ES, Piga M, Mangoni A, Passiu G, Gremese E, Ferraccioli G. Antimalarial use and arrhythmias in COVID-19 and rheumatic patients: a matter of dose and inflammation? Ann Rheum Dis. 2021 Mar;80(3):e29. doi: 10.1136/annrheumdis-2020-217828. Epub 2020 May 18. No abstract available. PMID 32424028
- [Derived] Erre GL, Piga M, Fedele AL, Mura S, Piras A, Cadoni ML, Cangemi I, Dessi M, Di Sante G, Tolusso B, Gremese E, Cauli A, Mangoni AA, Saba PS, Carru C, Ferraccioli G, Mathieu A, Passiu G. Prevalence and Determinants of Peripheral Microvascular Endothelial Dysfunction in Rheumatoid Arthritis Patients: A Multicenter Cross-Sectional Study. Mediators Inflamm. 2018 Feb 1;2018:6548715. doi: 10.1155/2018/6548715. eCollection 2018. PMID 29483841